CLINICAL TRIAL: NCT06324929
Title: Optimizing a Digital AEP Risk Intervention With Native Women and Communities
Acronym: CARRIINative
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: University of Minnesota (Other); Missouri Breaks Industries Research, Inc. (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Karen Ingersoll, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SBS6760; R61AA030581-01 (NIH)
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Exposed Pregnancy; Unplanned Pregnancy; Alcohol Use, Unspecified; Contraception Use; Sexual Behavior
Keywords: Native American; female; adult; contraception; alcohol; digital intervention; optimization; mHealth (mobile health)
MeSH Terms: conditions — Alcohol Drinking; Sexual Behavior

STUDY DESIGN:
Intervention Model Description: Mixed methods research during Aim 1 will include 4 different components. They are:
  1. Convene working group of Native American stakeholders.
  2. Collect data using a 35-minute survey of demographics, AEP risk, device use, recommendations for recruitment methods, and interest in subsequent trial with 300 Native women respondents, targeting approximately 100-150 per region
  3. Conduct Iterative prototyping of existing and proposed CARRII components with 60 Native women in 10 focus group discussions.
  4. Conduct User Testing of existing CARRII and candidate components with Think-Aloud methods among 20 Native women.
  In Aim 2, we will calculate baseline to 6-week improvements in knowledge about drinking and contraception, intention to change, self-efficacy and readiness for change, differences in drinking and contraception behaviors, and effect sizes of each component. The focus of this aim is to determine the effect size of each novel component.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aim 1 Survey (No Intervention): We will enroll up to 300 Native women ages 18-44 to complete a 35-minute survey to characterize demographics, parity, literacy, AEP risk, drinking levels, knowledge of FASD, location, Tribal affiliation, cultural preferences for tailoring, preferred digital platforms, methods of access to mobile devices/Internet, and interest in a digital women's health study about alcohol and birth control
- Rapid Pilot Testing (Experimental): Participants will complete a baseline past month TLFB (timeline follow-back) of alcohol use and contraception use during sex and a short online survey evaluating knowledge about AEP risk, intentions to change, self-efficacy for change, and readiness to change alcohol use and contraception behaviors. Each cohort of 10 participants will receive one of the 5 novel components (telephone-administered TLFB 2 weeks after study enrollment, mailed pregnancy test arriving 10-14 days after enrollment, digital safer sex and drink reduction skills training accessible across the 6-week period, automated texting prompting usage of skills across the 6-week period, or anonymized community message board across the 6-week period). Participants will complete a second TLFB for the past 6 weeks, and a short survey to rate the component they experienced, a System Usability Scale on their component, and measures of short-term knowledge, intentions to change, self-efficacy for change, and readiness to change.
  Interventions: Behavioral: CARRII Native Rapid Pilot Testing

INTERVENTIONS:
Behavioral: CARRII Native Rapid Pilot Testing — The candidates that will be tested are: 1) Telephone-administered 30 day timeline follow-back of drinking, sex, and contraception, administered by phone at enrollment and monthly, which should increase awareness of AEP risk and motivation for alcohol and contraception behavior change, 2) Mailed pregnancy tests sent monthly to raise consciousness of pregnancy risk and to detect a new pregnancy early, which should increase motivation for contraception behavior change, 3) Automated, personalized digital safer sex and drink counting/reduction skills training, to improve drinking self-management skills and self-efficacy for drinking reduction and contraception use, 4) Fully automated text messages prompting usage of safer sex and drink reduction skills, which should increase self-efficacy for behavior change, and 5) access to an anonymized Community Message Board of Native women to discuss challenges in behavior change, which should increase perceived social support.
  Arms: Rapid Pilot Testing

SUMMARY:
The purpose of Aim 1 of the study is to gather quantitative and qualitative information to inform the development of a digital app tailored for Native American women to help them avoid a pregnancy affected by alcohol. In Aim 2, we will Pilot test 5 new candidate components tailored to Native women at risk of AEP

DETAILED DESCRIPTION:
Alcohol exposed pregnancy (AEP) can result in Fetal Alcohol Spectrum Disorders (FASDs) that cause lifelong costly disabilities from brain, organ, tissue, and neurological damage. While over 3.3 million US women per month are at risk for AEP, risk for AEP among Native American (Native) women is higher, due to low contraception use and high binge drinking rates. For example, 20% of sexually active Native women in the Southwestern US are at risk for AEP, and 52% of pregnancies in the Navajo Nation are unplanned, compared to 45% nationally. Among pregnant women from Great Plains tribes, nearly 30% drink at binge levels and do not use contraception to prevent pregnancy. Among another sample of Native women from Great Plains tribes, 65% were sexually active, not seeking pregnancy, and not using contraception.

For Aim 1 we will implement four study methods to evaluate and tailor CARRII digital intervention components for Native women and prepare them to be used in a subsequent trial. These iterative mixed methods formative studies include:

1. Develop an ongoing Native Partners Working Group to review study plans and findings over time with the research team,
2. Collect quantitative surveys from Native women to estimate rates of AEP risk, interest/ ability to participate, health literacy, and other factors (n=300),
3. Conduct Focus Groups to prototype and tailor new CARRII components (up to n=60), and
4. Conduct Think-aloud User Testing (n=20) to finalize a draft of the CARRII Native intervention to prepare for development on a responsive design platform.

After incorporating input from participants (SA 1) and the Native Partners Working Group, we will pilot candidate components (SA2) to assess independent effects on AEP behavioral risk factors (drinking and contraception) while considering practical aspects such as frequency and duration of contact with participants, and costs of each component.

AEP can be prevented by avoiding an unintended pregnancy or reducing alcohol intake by those who may become pregnant. PI Ingersoll was a PI on the seminal CHOICES study that developed the first efficacious theory-based AEP intervention, with 4 Motivational Interviewing (MI) counseling sessions. PI Hanson adapted CHOICES for Native women in tribal communities. The Native-adapted CHOICES reduced AEP risk among Native women, but was too costly to sustain for high-risk women and communities.

In contrast, theory-based digital interventions are highly accessible, more convenient, scalable, and more sustainable, while still efficacious. In R34AA020853, Ingersoll piloted the first automated digital AEP intervention, CARRII. A nationwide pilot randomized controlled trial (RCT) showed that CARRII (but not the education control) significantly reduced AEP risk and pregnancy risk at 3 and 6 months, and drinking risk at 3 months. However, CARRII was studied among general population women, and not Native American women specifically.

Because rates of unintended pregnancy and binge drinking that create AEP risk are inequitable between Native women and the general population, CARRII will be tailored to and optimized for this priority subgroup. Guided by the Multiphase Optimization Strategy (MOST), we will tailor CARRII's existing components for Native women and systematically test proposed novel components (derived from formative work with Native women), to develop an efficient and scalable intervention tailored to Native women at risk of AEP. Optimizing CARRII for Native women will require measuring the efficacy and costs of components to find a balance between impact and affordability for Native communities. The overarching goal of this R61/R33 proposal is to determine the optimal combination of novel intervention strategies to include with CARRII (tailored for Native women) that maximizes digital intervention efficacy at feasible cost for Native communities. Achieving R61 milestones will permit progression to the R33 phase.

ELIGIBILITY:
Inclusion Criteria for survey:

* Native American

Inclusion Criteria for rapid pilot testing:

* Native American
* Risk for Alcohol Exposed Pregnancy

Exclusion Criteria:

-

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-09-19 (Estimated); Study Completion 2025-10-17 (Estimated)

PRIMARY OUTCOMES:
Rate of risky drinking | 6 weeks
  Defined as binge drinking, and/or drinking over daily risk levels. Unit of measure: Rate of risky drinking Measurement tool: TLFB (timeline follow-back) of alcohol use and contraception use during sex Outcomes 1 and 2 are combined to define alcohol-exposed pregnancy risk.
Rate of ineffective/absent contraception use | 6 weeks
  Defined per method used, or none, when having sex. Unit of measure: Rate of ineffective/absent contraception use Measurement tool: TLFB (timeline follow-back) of alcohol use and contraception use during sex Outcomes 1 and 2 are combined to define alcohol-exposed pregnancy risk.
Rate of AEP Risk | 6 weeks
  Combination of drinking above risk levels and inconsistent or absent use of effective contraception

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia Fontaine Research Park, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
We will comply with NIH data sharing protocols and will upload data to the NIAAA Data archive.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after data analysis is completed, we will deposit it in the data archive
Access Criteria: Other researchers can request data from the NIAAA Data Archive using their procedures.
URL: https://www.niaaa.nih.gov/research/niaaa-data-archive

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2025-03-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT06324929/Prot_SAP_002.pdf
  • Informed Consent Form: survey (2024-12-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT06324929/ICF_003.pdf
  • Informed Consent Form: rapid pilot testing (2024-12-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT06324929/ICF_004.pdf